CLINICAL TRIAL: NCT06197087
Title: Evaluation of Chronotype and Central Sensitization in Patients With Fibromyalgia Syndrome, Cross-sectional Study
Brief Title: Evaluation of Chronotype and Central Sensitization in Patients With Fibromyalgia Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oğuzhan Kandemir (Other)
Responsible Party: Sponsor-Investigator, Oğuzhan Kandemir, physical medicine and rehabilitation specialist doctor, Afyonkarahisar Health Sciences University
Organization: Afyonkarahisar Health Sciences University (Other)
Other Study IDs: chronotypeandfibromyalgia2023
Record Dates: First submitted 2023-12-10; First posted 2024-01-09 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Chronotype; Fibromyalgia Syndrome
Keywords: fibromyalgia syndrome; Chronotype; central sensitization; disability; quality of life
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: cross-sectional observational survey study — Patients' pain intensity (with VAS), quality of life (with SF-12), sleep quality (with Pittsburgh sleep quality scale), anxiety and depression symptoms (with Beck Depression Inventory), cognitive aspect of pain (with Pain Catastrophizing Scale), presence of central sensitization (with the central sensitization scale), functional status (with the Fibromyalgia impact questionnaire), and chronotype preferences will be evaluated with the Morningness and Eveningness Questionnaire.

SUMMARY:
The aim of study is to examine the chronotype preferences of patients with fibromyalgia syndrome and the relationship between central sensitization and chronotype, and to examine its relationship with pain intensity, disability and quality of life.

DETAILED DESCRIPTION:
Fibromyalgia Syndrome (FMS); It is a syndrome characterized by chronic pain occurring in more than one part of the body and accompanied by fatigue, sleep disturbance, impairment in quality of life and daily functionality. Although FMS is seen in different age groups, it is most common in middle-aged women. FMS is classified as central sensitization syndrome, in which there is an abnormal response to painful stimuli and the processing of nociceptive stimuli in the central nervous system. In patients with FMS, pain may cause sleep disturbances such as non-restorative sleep or difficulty initiating or maintaining sleep. It is estimated that 65-99% of patients with FMS experience sleep disorders. Circadian rhythms reflect 24-hour physiological and behavioral cycles within each individual. Based on individual differences in the timing of these innate rhythms, individuals can be divided into 3 phenotypes (i.e., chronotypes): morning type (M-highest level of alertness in the morning), evening type (E most active in the evening), and intermediate type (I-neither M nor E). Chronotype is explained by both genetic and environmental factors and can be considered a fairly robust trait throughout adulthood. A study assessing 1548 people with FMS with an online survey including questions about sleep quality, well-being, pain, chronotype and FMS impact shows that late chronotypes are more affected by fibromyalgia. In another study conducted in 2019, patients with FMS were grouped according to chronotype preferences and showed that there was a strong relationship between FMS severity and poor quality of life in evening individuals.

The aim of study is to examine the chronotype preferences of patients with fibromyalgia syndrome and the relationship between central sensitization and chronotype, and to examine its relationship with pain intensity, disability and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed according to ACR 2016 Fibromyalgia Syndrome Diagnostic criteria Continuing complaints for at least 3 months

Exclusion Criteria:

* Neurological and Inflammatory diseases Pregnancy Malignancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients who applied to Yerköy State Hospital Physical Medicine and Rehabilitation Polyclinic and Afyonkarahisar Health Sciences University Faculty of Medicine Hospital Physical Medicine and Rehabilitation Polyclinic and were followed up with the diagnosis of FMS for at least 3 months will be included in the study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Central Sensitization Inventory | 1 hour
  Central Sensitization Inventory (CSI) The CSI is a two-part questionnaire that contains a 25-item survey (Part A) that assesses the frequency of health-related symptoms associated with central sensitivity syndromes and a brief survey (Part B) asking if patients have been diagnosed with specific disorders (Neblett et al., 2013). For the purposes of this study, only responses from the 25-item survey were included. Participants are asked to rate each question on a 5-point scale with 0 meaning "never" and 4 meaning "always." A summed response is obtained with a total possible score of 100. Higher CSI scores represent greater self-reported symptomology. A cutoff score of 40 or greater has shown acceptable psychometrics for identifying patients with central sensitivity syndromes
Morning and Evening Survey | 1 hour
  Sleep is one of the most commonly used tools to assess chronotype preferences. This screening questionnaire, consisting of 19 items, has a rating range between 16 and 86. Scoring results were classified as follows: evening types scoring between 16 and 41, morning types scoring between 59 and 86, and no types scoring between 42 and 58. The Turkish version has been shown to have good validity and reliability.
Fibromyalgia Impact Survey | 1 hour
  It was developed by Burckhardt and his colleagues in 1991. It is the most commonly used scale to evaluate functional status in patients with FMS. It evaluates 10 different characteristics, including physical functioning, well-being, missed work days, difficulty at work, pain, fatigue, morning fatigue, stiffness, anxiety and depression. The total score varies between 0 and 80. A high score indicates that the disease affects the person more. Cronbach's alpha coefficient for all items was 0.73.

SECONDARY OUTCOMES:
VAS | 1 hour
  Visual Pain Scale (VAS), which is easy to understand, apply and interpret and provides valid and reliable data in a short time, is the most used method in clinics. Using a 100 mm visual linear scale, the patient is told that at point 0 there is no pain, and at point 100 it is the most severe pain ever felt in life, and the patient is asked to place a mark on the point corresponding to his pain.
Pittsburg Sleep Quality Index (PSQI) | 1 hour
  The first 18 questions answered by the participant are used in calculating the PSQI total score and component scores. The 18 questions answered by the participant included sleep quality (component 1), sleep latency (component 2), sleep duration (component 3), habitual sleep efficiency (component 4), sleep disturbance (component 5), sleep medication use (component 6), and It provides information about 7 components, including daytime sleep dysfunction (component 7). Each component is evaluated on a scale of 0-3 points. The sum of these 7 component scores gives the total PSQI score. The total PSQI score varies between 0-21. While the sleep quality of individuals with a total score of 5 or less is considered "good", the sleep quality of individuals with a score above 5 is considered "bad".
Beck Depression Anxiety Scale | 1 hour
  Beck Depression Inventory is a self-rating scale consisting of 21 items. Each item was given a score between 0 and 3, the highest score that could be obtained from the scale was 63 and the lowest score was 0. A high score from the scale indicates that the severity or level of depression is high.
Pain Catastrophizing Scale | 1 hour
  Sullivan et al. It is a 13-item self-report inventory using a 5-point Likert scale (0-4) developed by To measure the extent to which people catastrophize in response to pain. The original scale consists of three sub-factors called helplessness, magnification and rumination.
SF-12 | 1 hour
  SF-12 is an easy-to-administer survey with proven reliability and validity, obtained by shortening and simplifying the SF-36. It is used to evaluate physical and mental health, the two main components of general health status. Consisting of twelve questions, SF-12 has mental and physical component scores. High scores indicate good health.

CONTACTS AND LOCATIONS:
Overall Officials: sevda adar, Principal Investigator — Afyonkarahisar Health Sciences University; ümit dündar, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrade A, Vilarino GT, Sieczkowska SM, Coimbra DR, Bevilacqua GG, Steffens RAK. The relationship between sleep quality and fibromyalgia symptoms. J Health Psychol. 2020 Aug;25(9):1176-1186. doi: 10.1177/1359105317751615. Epub 2018 Jan 8. PMID 29310453
- [Background] Boomershine CS. Fibromyalgia: the prototypical central sensitivity syndrome. Curr Rheumatol Rev. 2015;11(2):131-45. doi: 10.2174/1573397111666150619095007. PMID 26088213
- [Background] Fitzcharles MA, Ste-Marie PA, Goldenberg DL, Pereira JX, Abbey S, Choiniere M, Ko G, Moulin DE, Panopalis P, Proulx J, Shir Y; National Fibromyalgia Guideline Advisory Panel. 2012 Canadian Guidelines for the diagnosis and management of fibromyalgia syndrome: executive summary. Pain Res Manag. 2013 May-Jun;18(3):119-26. doi: 10.1155/2013/918216. PMID 23748251
- [Background] Theadom A, Cropley M, Humphrey KL. Exploring the role of sleep and coping in quality of life in fibromyalgia. J Psychosom Res. 2007 Feb;62(2):145-51. doi: 10.1016/j.jpsychores.2006.09.013. PMID 17270572
- [Background] Turkoglu G, Selvi Y. The relationship between chronotype, sleep disturbance, severity of fibromyalgia, and quality of life in patients with fibromyalgia. Chronobiol Int. 2020 Jan;37(1):68-81. doi: 10.1080/07420528.2019.1684314. Epub 2019 Nov 5. PMID 31687843
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783
- [Background] Czeisler CA, Gooley JJ. Sleep and circadian rhythms in humans. Cold Spring Harb Symp Quant Biol. 2007;72:579-97. doi: 10.1101/sqb.2007.72.064. PMID 18419318
- [Background] Barclay NL, Rowe R, O'Leary R, Bream D, Gregory AM. Longitudinal Stability of Genetic and Environmental Influences on the Association between Diurnal Preference and Sleep Quality in Young Adult Twins and Siblings. J Biol Rhythms. 2016 Aug;31(4):375-86. doi: 10.1177/0748730416653533. Epub 2016 Jun 23. PMID 27339174